CLINICAL TRIAL: NCT01866462
Title: A Pilot Study of the Effect of NM-504 Cobiotic Formulation on the Efficacy and Tolerability of Metformin in Patients With Metformin Intolerance
Brief Title: Pilot Study of the Effect of MN-504 Cobiotic Formulation on the Efficacy and Tolerability of Metformin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NuMe Health (Industry)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ProCo Metformin
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin, NM504 (Experimental): metformin 500mg b.i.d. with NM504 b.i.d. for 1 week followed by metformin 500mg t.i.d. with NM504 b.i.d. for 1 week.
  Interventions: Other: NM504
- Metformin, Placebo (Placebo Comparator): metformin 500mg b.i.d. with Placebo b.i.d. for 1 week followed by metformin 500mg t.i.d. with Placebo b.i.d. for 1 week.

INTERVENTIONS:
Other: NM504 — NM504 is a medical food designed to shift the dysbiota reported in type 2 diabetes. The placebo is carboxymethylcellulose prepared to look, taste and mix like NM504.
  Other Names: NM-504; NM-504 cobiotic; NM-504 cobiotic formula; NM504 cobiotic; NM504 cobiotic formula
  Arms: Metformin, NM504

SUMMARY:
The purpose of the study is to determine if NM504 will prevent GI side effects that are associated with using metformin for the treatment of diabetes.

DETAILED DESCRIPTION:
Only subjects with known intolerance to metformin will be recruited and enrolled in this study. When a participant qualifies, after signing the consent, they will be asked to complete a questionnaire about medical history which will be reviewed with the coordinator. Their height, weight, and blood pressure will be measured, and their medications will be reviewed. They will be taught how to measure their fasting blood glucose by a finger stick. They will be given metformin and asked to take a 500mg tablet twice day before breakfast and dinner starting the next day with breakfast. They will be given doses of NM504 or a placebo in a pouch to be mixed with 6 ounces of water before breakfast and dinner as a smoothie drink starting before breakfast the next day. Before consuming the first smoothie each day and before eating any food each day they will be asked to record their fasting finger stick blood glucose and complete the questionnaire about their bowel habits. The study takes place in two-week segments with a two week washout in between. They will receive metformin in both periods, but they will receive NM504 during one 2-week segment and a placebo smoothie during the other two-week segment. Five subjects will receive NM504 and 5 subjects will be assigned placebo during the initial 2 weeks. The treatment sequence will be randomly assigned. After the 2 week washout period the subjects will cross over to either placebo or NM504.

Phone Visit 1: week 1 subjects will receive a call from the coordinator to see how they are tolerating the metformin and the smoothies. An increase in metformin dose to 500mg 3 times a day may or may not happen.

Clinic Visit 2: week 2, Subjects will bring bottle of metformin and empty packages of smoothie powder to the visit along with logs of their daily fasting finger stick blood glucose and their daily bowel questionnaires. Their body weight weight will be measured.

Clinic Visit 3: week 4, subjects will be asked about their metformin tolerance and body weight will be measured. They will be given metformin and asked to take a 500 mg pill twice a day before breakfast and dinner starting the next day before breakfast. Before consuming the first smoothie each day, and before eating any food each day, subjects will be asked to record a fasting finger stick blood glucose and complete the questionnaire about bowel habits.

Phone Visit 2: week 5 subjects will be asked about their tolerance to metformin and the smoothies. They may or may not be asked to increase their 500mg dose of metformin from 2 times a day to 3 times a day.

Clinic Visit 4: week 6, Subjects will bring the bottle of metformin and the empty packages of the smoothie powder to the visit along with the logs of daily fasting finger stick blood glucose and daily bowel questionnaires. Their body weight will be measured at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or a female with type 2 diabetes
* Known tolerance to metformin
* 18 years of age or older
* Body mass index that is not less than 20 kg/m2

Exclusion Criteria:

* Not pregnant or breast feeding a baby.
* Not taking chronic medication that has not had a stable dose for 1 month or longer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Metformin Tolerance | 6 Weeks
  Fecal frequency, fecal consistency, fecal score and incidence of diarrhea will be assessed using the validated King's Stool Chart.

SECONDARY OUTCOMES:
Fasting Blood Glucose | 6 weeks
  Fasting blood glucose will be measured by finger stick daily.
GI Symptoms | 6 weeks
  Other possible GI symptoms such as sensations of bloating and flatulence will be measured with a questionnaire adapted from the validated Irritable Bowel Syndrome Global Improvement Scale.
GI Stool Profile | 6 weeks
  Stool will be collected at baseline, after the initial 2 week treatment, at the end of the washout period, and at the completion of the study. The complete stool GI function profile assessed by Genova Diagnostics will be performed.
Weight Loss | 6 weeks
  Body weight will be measured at each clinic visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States